CLINICAL TRIAL: NCT02605707
Title: Autologous Endothelial Progenitor Cells Transplantation for Chronic Ischemic Stroke
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Southern Medical University, China (Other)
Collaborators: Second Affiliated Hospital of Guangzhou Medical University (Other)
Responsible Party: Principal Investigator, Zhen-Zhou Chen, Department of Neurosurgery, Zhujiang Hospital, Southern Medical University, China
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2011Y1-00033-6
Record Dates: First submitted 2015-11-12; First posted 2015-11-16 (Estimated); Last update posted 2021-04-02 (Actual); Status verified 2021-04

CONDITIONS: Stroke
Keywords: Endothelial Progenitor Cells; Transplantation; Stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intravenous stem cell transplantation (Experimental): Intravenous transplantation of autologous endothelial progenitor cells plus conventional treatment include rehabilitation
  Interventions: Drug: Intravenous stem cell transplantation
- Conventional treatment (No Intervention): Control group receive conventional stroke treatment that include rehabilitation

INTERVENTIONS:
Drug: Intravenous stem cell transplantation — Intravenous injection of autologous endothelial progenitor cells transplantation
  Arms: Intravenous stem cell transplantation

SUMMARY:
Stroke is a frequently occurring and common diseases in nervous system,and most of the survivors will remain disorders of motor,sensory and cognition function.Stem cell transplantation provides a promising approach for rehabilitation. The main objective of this study is to evaluate the efficacy and safy of the transplantation of autologous endothelial progenitor cells in patients with chronic stroke.

DETAILED DESCRIPTION:
Stroke is a frequently occurring and common diseases in nervous system,and most of the survivors will remain disorders of motor,sensory and cognition function.It will brought heavy burden to patients themselves,their family and society.Drugs,rehabilitation excise and hyperbaric oxygen will improve functions after acute stroke.However,in the chronic ischemic stroke,there was few methods to improve the functions.In recently research,stem cell will be a new methods to improve the neural function after through differentiate to nervous cells and secrete some neurotrophic factors to repair the damage. In this study, the investigators will assess the safety and feasibility of intracerebral transplantation of autologous endothelial progenitor cells in patients with chronic ischemic stroke. The neurological outcome will be determined after transplantation.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18-80 chronic ischemia stroke or patients
* With stroke history of more than 6 months, less than 60 months
* NIHSS (NIH stroke scale) score of 7 or more points
* Internal carotid artery territory infarction measured by MRI
* Can be hospitalized and signed informed consent
* With fewer effect by traditional post-stroke treatments or rehabilitations

Exclusion Criteria:

* Lacunar infarction
* Recurrent thrombotic diseases less than 6 months
* Hemorrhage stroke,brain tumor or MRI show the occlusion is not in the middle cerebral artery territory
* Pregnant women
* Can't tolerate the test because of other disease, such as heart failure, liver failure, renal failure, abnormal blood coagulation, AIDS, combine other tumor or special condition
* Penicillin anaphylaxis or some other drugs allergy
* Autoimmune disease
* Inaccessibility for follow up

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2014-11; Primary Completion 2017-12 (Actual); Study Completion 2020-02 (Actual)

PRIMARY OUTCOMES:
Change from baseline in Fugl-Meyer Scale at 24 months | 1,3,6,12 and 24months

SECONDARY OUTCOMES:
Change from baseline in NIH Stroke Scale at 24 months | 1,3,6,12 and 24months
Change from baseline in Barthel Index at 24 months | 1,3,6,12 and 24months
Change from baseline in SSS at 24 months | 1,3,6,12 and 24months
Change from baseline in mRS at 24 months | 1,3,6,12 and 24months
Improvement of vision measured by brain visual examination | 1,3,6,12 and 24months

CONTACTS AND LOCATIONS:
Overall Officials: ZhenZhou Chen, MD, phD, Principal Investigator — Department of Neurosurgery, Zhujiang Hospital
Locations (1):
- Zhujiang Hospital, Southern Medical University, Guangzhou, Guangdong, China